CLINICAL TRIAL: NCT01168180
Title: Efficacy of Traditional Thai Massage on Patients With Scapulocostal Syndrome
Brief Title: Traditional Thai Massage and Scapulocostal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Assoc Prof. Dr. Wichai Eungpinithpong, Faculty of Associated Medical Sciences, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 527090004-4
Record Dates: First submitted 2010-07-19; First posted 2010-07-23 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2011-06

CONDITIONS: Scapulocostal Syndrome
Keywords: Traditional Thai Massage; Scapulocostal Syndrome
MeSH Terms: interventions — Medicine, Thai Traditional; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Thai massage (Experimental): The participants will receive thirty minutes session of traditional Thai massage onto the scapular region for 9 sessions over a period of 3 weeks
  Interventions: Other: Traditional Thai massage
- Ultrasound therapy and hot pack (Active Comparator): The participants will receive thirty minutes session of Ultrasound therapy and hot pack for 9 sessions over a period of 3 weeks
  Interventions: Other: Ultrasound therapy and hot pack

INTERVENTIONS:
Other: Traditional Thai massage — The participants will receive thirty minutes session of traditional Thai massage onto the scapular region for 9 sessions over a period of 3 weeks
  Arms: Traditional Thai massage
Other: Ultrasound therapy and hot pack
  Arms: Ultrasound therapy and hot pack

SUMMARY:
The purpose of this study is to evaluate the efficacy of traditional Thai massage on pain intensity, pressure pain threshold, muscle tension, anxiety, cervical range of motion, patient satisfaction and side effects in the treatment of scapulocostal syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age between 18 - 50 years old
3. The participants have experienced spontaneous scapular pain (VAS ≥ 3) for longer than 12 weeks (chronic) and that at least one trigger point will be present in the scapular region (serratus posterior superior, rhomboid groups, levator scapulae and trapezius muscles). Trigger points will be diagnosed as the presence of focal tenderness in a taut band and with pain recognition.
4. The participants will be able to follow instructions.
5. Good communication and cooperation.

Exclusion Criteria:

1. A history of the following diseases or disorders:

   * Rotator cuff disease
   * Cervical radiculopathy
   * Degenerative shoulder joint disease
   * Shoulder stiffness
2. Contraindications of traditional Thai massage

   * Contagious skin disease
   * Injury or inflammation of muscle
   * Bone fracture and/or joint dislocation
   * Open wound
   * Uncontrolled hypertension
   * Drug and/or alcohol intoxication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity (Visual analog scale) | 4 months
  The intensity of pain will be reported by the participant on a numerical analog scale ranging from 0 to 10. Zero indicates no pain anywhere and 10 indicates the most pain ever experienced.

SECONDARY OUTCOMES:
Pressure Pain Threshold | 4 months
Muscle tension (Visual analog scale) | 4 months
State Anxiety Inventory | 4 months
patient satisfaction | 3 weeks
Side effects | 3 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Associated Medical Sciences, Khon Kaen University, Muang, Changwat Khon Kaen
  - School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Muang, Changwat Khon Kaen